CLINICAL TRIAL: NCT01618526
Title: ButCoIns GUTS: - Gut Immunological Effects of Resistant Starch and Arabinoxylans in Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: V02062012
Record Dates: First submitted 2012-05-30; First posted 2012-06-13 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2013-08

CONDITIONS: Metabolic Syndrome
Keywords: Dietary fibers; Butyrate; Short Chain Fatty Acids; Colon; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Carbohydrate Diet (Active Comparator): 4 weeks of intervention with a diet rich in Arabinoxylans and Resistent Starch
  Interventions: Dietary Supplement: Healthy Carbohydrate Diet
- Western Style Diet (Placebo Comparator): 4 weeks of intervention with a diet with low content of Resistent Starch and Arabinoxylans.
  Interventions: Dietary Supplement: Western Style Diet

INTERVENTIONS:
Dietary Supplement: Western Style Diet — Cross over design with two intervention diet: Healthy Carbohydrate Diet with approximally 55 grams of dietary fibers (Arabinoxylans and Resist Starch) compared with a Western Style Diet with a low content of dietary fibers.
  Arms: Western Style Diet
Dietary Supplement: Healthy Carbohydrate Diet — Cross over design with two intervention diet: Healthy Carbohydrate Diet with approximally 55 grams of dietary fibers ( Arabinoxylans and Resistent Starch) compared with Western Style Diet with low content of dietary fibers
  Arms: Healthy Carbohydrate Diet

SUMMARY:
Dietary fibers including resistent starch, RS, and arabinoxylans, AX, have been shown to have anti-inflammatory effects and to change the composition of the faecal micro flora in the colon.

In this unblinded dietary intervention cross-over study 20 subjects with metabolic syndrome are randomized to two types of diet intervention: a low and a high fiber diet. The participants are subjected to endoscopy before and in the end of each intervention.

DETAILED DESCRIPTION:
Dietary fibers including resistent starch, RS, and arabinoxylans, AX, have been shown to have anti-inflammatory effects and to change the composition of the faecal micro flora in the colon.

In this unblinded dietary intervention cross-over study 20 subjects with metabolic syndrome are subjected to two types of diet intervention:

1. a western style diet, WSD, with a low fiber content and
2. a healthy carbohydrate diet, HCD, a high fiber diet. Between the two 4-weeks diet is a wash-out period of four to eight weeks. The participants are subjected to endoscopy with tissue samples before and in the end of each intervention. Fecal and blood samples will be collected at the same time.

We hypothesize that a high content of resistent starch and arabinoxylans increases colonic butyrate concentration, changes colon's mucosal immune system and the microbiota.

A small pilot study will be carried out on 12 healthy volunteers in order to obtain a reference to participants with metabolic syndrome. The healthy volunteers will be subjected to an endoscopy but no dietary intervention.

ELIGIBILITY:
Inclusion Criteria: At least 3 out of 5 following criteria:

* Central obesity (Female > 80 cm, Male > 94 cm)
* HDL cholesterol (Female < 1,03 mmol/L, Male < 1,29 mmol/L)
* Bloodpressure (> 130/85 mmHg)
* Fasting Blood Glucose > 5,6 mmol/L

Exclusion Criteria:

* Diabetes
* Gastrointestinal disease
* Serious liver, heart or kidney disease
* Anticoagulation treatment
* Anaemia
* Corticosteroid treatment
* Waist circumference above 130 cm
* Alcohol or drug addiction
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feces-short chain fatty acids | Baseline and 4 weeks
  Concentration of short chain fatty acids

SECONDARY OUTCOMES:
A change in gut microbiome evaluated by 16 S-RNA analysis | Baseline and 4 weeks
Change in Nuclear Factor-kappa B (NF-кB) described by gene expression analysis. | Baseline and 4 weeks
Change in production of pro inflammatory cytokines on mucosal level (IFN-γ, TNF-α, IL-17). | Baseline and 4 weeks
Change in production of regulatory cytokines on mucosal level and in peripheral blood mononuclear cell (IL-22, IL-10 TNF-β). | Baseline and 4 weeks
Activation of T-cells in mucosa described by reduced expression of CD25 and CD69. | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Knud Erik Bach Knudsen, Professor, Principal Investigator — Aarhus University, Department of Animal Sciens
Locations (1):
- Aarhus University, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Hald S, Schioldan AG, Moore ME, Dige A, Laerke HN, Agnholt J, Bach Knudsen KE, Hermansen K, Marco ML, Gregersen S, Dahlerup JF. Effects of Arabinoxylan and Resistant Starch on Intestinal Microbiota and Short-Chain Fatty Acids in Subjects with Metabolic Syndrome: A Randomised Crossover Study. PLoS One. 2016 Jul 19;11(7):e0159223. doi: 10.1371/journal.pone.0159223. eCollection 2016. PMID 27434092